CLINICAL TRIAL: NCT05390047
Title: The International Subcutaneous Implantable Cardioverter Defibrillator Registry (iSuSi)
Acronym: iSuSI
Status: Recruiting | Type: Observational
Sponsor: University of Luebeck (Other)
Collaborators: Prof. Jürgen Kuschyk, M.D (Unknown); Giovanni Forleo, M.D. (Unknown); Mauro Biffi, M.D. (Unknown)
Responsible Party: Principal Investigator, Prof. Roland Richard Tilz, Prof. Dr. med. Roland Richard Tilz, University of Luebeck
Other Study IDs: ISuSI 1.0
Record Dates: First submitted 2022-02-22; First posted 2022-05-25 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Sudden Cardiac Death
Keywords: subcutaneous implantable cardioverter defibrillator
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The entirely subcutaneous implantable defibrillator (S-ICD) (Emblem, Boston Scientific, Marlborough, MA, USA) was introduced as a new therapeutic alternative to the conventional transvenous ICD in 2009 and implantations are rapidly expanding since then.1 Implantation of the S-ICD seems to reduce implant-related perioperative complications such as pneumothorax, hematoma and cardiac tamponade.

The aim of this multicenter registry is thus to assess the outcome of patients following an S-ICD implantation in a real-world setting.

DETAILED DESCRIPTION:
The S-ICD has a CE mark and is FDA approved since 2012 and is mentioned as a potential therapy strategy in the current AHA guidelines on the management of patients with ventricular arrhythmias.2 However, although implant-related complications seem to be reduced by the S-ICD in randomized controlled trials, the rate of inappropriate shocks remains high in S-ICD patients (10-13%).3-5 The most common reason for inappropriate shocks is cardiac oversensing, mostly due to T-wave oversensing or low amplitude of the subcutaneous signal, which not commonly found in patients with transvenous ICDs. Data on the role of the Defibrillation Threshold Testing (DFT), the rate of infectious complications (lead or device complications), the use of the S-ICD in children and adolescents, and the outcome of patients with an S-ICD according to their underlying cardiac substrate are sparse. The aim of this multicenter registry is thus to assess the outcome of patients following an S-ICD implantation in a real-world setting with a special focus on perioperative complication rate, the role of DFT testing in S-ICD, the use of the S-ICD in cohorts that are underrepresented in clinical studies (adolescents and geriatrics), the outcome and risk factors of ineffective, inappropriate and appropriate shocks and the differences in outcomes according to the underlying cardiac disease.

ELIGIBILITY:
Inclusion Criteria:

* Implantation of an S-ICD, regardless of the technique
* At least 1 month of follow up
* At least 1 post-implantation assessment, in accordance to the routine clinical practice of every center (e.g. in person visit or remote follow up)

Exclusion Criteria:

- none

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in whom a S-ICD was implanted for primary or secondary prevention
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall complication rate | through study completion, an average of 2 years
  combination of device related complications and inappropriate shocks
Rate of appropriate shocks | through study completion, an average of 2 years
  Appropriate therapies delivered by the devices
Rate of inappropriate shocks | through study completion, an average of 2 years
  Inappropriate therapies delivered by the devices

SECONDARY OUTCOMES:
Device-related complication rate | immediately after the intervention/procedure/surgery"
  Rate of complications pertaining to the device
DFT impact | 2 year
  Impact of defibrillator function test (DFT) on long term arrhythmia outcome or mortality
Rate of replacements | 2 year
  Generator replacements
Role of Gender in primary outcomes | through study completion, an average of 2 year
  Analysis of the potential role of gender on the primary outcomes
Rate of device upgrades | through study completion, an average of 2 year
  need for device upgrade due to pacing needs

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for Rhythmology, Lübeck, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: Undecided